CLINICAL TRIAL: NCT00862498
Title: Examining Written Disclosure as an Intervention for Posttraumatic Stress Disorder
Brief Title: Examining Written Disclosure as a Treatment for Post-Traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Denise M. Sloan, Professor of Psychiatry, Boston University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-27236; R34MH077658 (NIH)
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; Written Disclosure; Written Emotional Disclosure; Narrative Exposure; Narrative Writing; Motor Vehicle Accident
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 Treatment in Clinic (Experimental): Participants will complete the written disclosure treatment in a clinic setting.
  Interventions: Other: Written Disclosure
- Group 2 Treatment via telephone (Experimental): Participants will complete the written disclosure treatment in their homes via telephone.
  Interventions: Other: Written Disclosure
- Group 3 Waitlist (No Intervention): Individuals will be placed on a waitlist for a period of 4 months, during which they will receive a phone call every other week to assess their suicidal ideation and post-traumatic stress disorder symptom severity.

INTERVENTIONS:
Other: Written Disclosure — Five sessions, each spaced 1 week apart, during which participants are asked to write about their motor vehicle accident for 30 minutes. The first session of the intervention also involves a description of common reactions to a motor vehicle accident and the rationale for this treatment.
  Other Names: Written Emotional Disclosure; Narrative Writing; Narrative Exposure
  Arms: Group 1 Treatment in Clinic; Group 2 Treatment via telephone

SUMMARY:
This study will test the effectiveness of writing about a traumatic incident to treat post-traumatic stress disorder in people who have been in car accidents.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is a chronic and debilitating disorder caused by experiencing a stressful or traumatic event. Although there is evidence that treatments for PTSD are effective, many people do not seek treatment or seek treatment only after their PTSD has become severe. This study will test a low-cost, brief, and easily implemented treatment that may encourage people to seek treatment for PTSD. The treatment, called written disclosure (WD), involves writing about the traumatic event that caused a person's PTSD. In this study, people who have PTSD as the result of a motor vehicle accident will test two versions of WD, one administered in a clinic and the other administered over the phone.

Participation in this study will last 5 weeks, with follow-up assessments continuing until 6 months after treatment. After screening, participants will be assigned to one of three conditions: WD treatment delivered in the clinic, WD treatment delivered via phone, and waitlist. The WD treatment involves five weekly writing sessions. During the first session, trauma reactions and the rationale for WD will be explained to all participants, and then participants will write for 30 minutes about their motor vehicle accident. The next four sessions will involve only writing for 30 minutes. For those receiving treatment in the clinic, a therapist will communicate directions and explanations to participants, and participants will have their heart rate activity recorded continuously for 5 minutes prior to writing and during the 30 minutes of writing. For those receiving treatment over the phone, explanations of the study will be provided in writing, and a study staff member will call participants before and after each writing session to ensure that participants understand the directions and are not experiencing any unexpected negative reactions after writing. Participants in the waitlist condition will not receive treatment for the first 4 months. After that period, they will be offered the WD treatment.

Assessments of all participants will occur at baseline, after treatment, and 3 months after treatment. Participants assigned to receive WD treatment, either in a clinic or via phone, will also be assessed 6 months after treatment. Assessments administered at these points will involve semi-structured clinical interviews, self-report questionnaires, and measures of mood-related symptoms. Participants receiving treatment will also complete self-report measurements of emotional response after each writing session and the Daily Experiences Questionnaire every day during the 5 weeks of treatment. Participants on the waitlist will also undergo assessments of suicidal thoughts and PTSD symptoms every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of post-traumatic stress disorder
* Involved in motor vehicle accident that occurred at least 3 months ago

Exclusion Criteria:

* Current diagnosis of mania, hypomania, bipolar depression, psychotic disorder, substance abuse disorder, or severe depression
* History of psychosis
* Active suicidality or history of two or more suicide gestures or attempts in the past year
* Significant cognitive impairment
* Current participation in a psychosocial treatment, such as individual or group therapy led by a clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Clinician-Administered Posttraumatic Stress Disorder Scale | Measured at baseline, post-treatment, and at 3- and 6-month follow-ups

SECONDARY OUTCOMES:
Beck Depression Inventory - Second Edition | Measured at baseline, post-treatment, and at 3- and 6-month follow-ups
Posttraumatic Cognitions Inventory | Measured at baseline, post-treatment, and at 3- and 6-month follow-ups
Anxious Driving Questionnaire | Measured at baseline, post-treatment, and at 3- and 6-month follow-ups
Client Satisfaction Questionnaire | Measured at the end of the last treatment session
Daily Experiences Questionnaire | Measured every day during the 5-week treatment period
Oswestry Disability Index | Measured at baseline, post-treatment, and at 3- and 6-month follow-ups
Quality of Life Inventory | Measured at baseline, post-treatment, and at 3- and 6-month follow-ups
Self-Assessment Manikin | Measured after each writing session
Last Day of Writing Questionnaire | Measured after the last writing session
Follow-Up Writing Questionnaire | Measured after the 3-month follow-up assessment
Alcohol Use Disorders Identification Test | Measured at baseline, post-treatment, and at 3- and 6-month follow-ups
Posttraumatic Stress Disorder Checklist - Civilian Version | Measured at baseline, post-treatment, and at 3- and 6-month follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Denise M. Sloan, PhD, Principal Investigator — VA Boston Healthcare System, National Center for PTSD; Boston University School of Medicine
Locations (1):
- VA Boston Healthcare System, National Center for PTSD, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sloan DM, Marx BP, Bovin MJ, Feinstein BA, Gallagher MW. Written exposure as an intervention for PTSD: a randomized clinical trial with motor vehicle accident survivors. Behav Res Ther. 2012 Oct;50(10):627-35. doi: 10.1016/j.brat.2012.07.001. Epub 2012 Jul 20. PMID 22863540